CLINICAL TRIAL: NCT07173205
Title: R00 Full Factorial Trial: Optimizing ASCENT
Brief Title: Optimizing the AYA Survivors' Coping and Emotional Needs Toolkit
Acronym: ASCENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Karly M Murphy, PhD, Principal Investigator, East Carolina University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-001496; R00CA248701 (NIH)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Depression; Cancer; Adolescent; Young Adult; Adult
Keywords: AYA; Adolescent and Young Adult; Cancer Survivorship; Depressive Symptoms; Digital Mental Health; Multiphase Optimization Strategy; Full Factorial Trial
MeSH Terms: conditions — Depression; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 2 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 3 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 4 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 5 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 6 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 7 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 8 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness)
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 9 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 10 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 11 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 12 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 13 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 14 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs); Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness).
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 15 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance)
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)
- Condition 16 (Experimental): Feeling component of ASCENT (psychoeducation about AYA cancer survivorship and depression); Doing component of ASCENT (an adaptation of behavioral activation that aims to help AYAs engage in enjoyable activities, achieve their goals, and live in accordance with their values); Thinking component of ASCENT (an adaptation of cognitive restructuring that aims to help AYAs identify, evaluate, and restructure their negative automatic thoughts and core beliefs); Being component of ASCENT (an adaptation of mindfulness training that aims to help AYAs maintain contact with the present moment with an attitude of acceptance); and Positivity component of ASCENT (an adaptation of a suite of evidence-based positive psychology interventions that aims to help AYAs savor the good things in life, use their strengths, and practice gratitude and kindness)
  Interventions: Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT)

INTERVENTIONS:
Behavioral: AYA Survivors Coping and Emotional Needs Toolkit (ASCENT) — Participants will receive access to a digital depression self-management tool (ASCENT), which aims to help AYAs manage symptoms of depression post-treatment. All users will have access to the core tool which includes daily mood tracking and a psychoeducational module about cancer and depression. Depending on assigned condition, participants will also receive access to up to 4 intervention modules which have been adapted from existing evidence-based treatments for digital delivery to AYAs through a rigorous user-centered design process. Within each module there are 6 micro-lessons that include an educational video, a real story from an AYA that demonstrates the topic, multiple choice questions that ask the participant to apply the educational information to the AYA story, open-ended questions that ask the participant to apply the educational information to their own experience, and a practice activity in which they are asked to try out a relevant skill.

SUMMARY:
Our team has developed a digital intervention that aims to help adolescent and young adult cancer survivors (AYAs) manage symptoms of depression. This tool includes one psychoeducation component and four components that are based on evidence-based interventions for depression. The goal of this study is to test which component or combination of components meaningfully contribute to improvements in depressive symptoms among AYAs.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment (adolescents 15-17, emerging adults 18-25, young adults 26-39)
* Age at diagnosis (adolescents 12-17, emerging adults 15-25, young adults 15-39)
* Time since completion of treatment: 1 month to 5 years
* Language: Fluent in English (spoken and written)
* Technology: Own smart phone with data plan

Exclusion Criteria:

* Mental Health: Current diagnosis of severe or persistent mental illness
* Suicidality: Severe suicidal ideation (including plan and intent)

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive Symptoms during Intervention Period | Baseline to Week 6
  The primary outcome for this study is change in depressive symptoms from Baseline to Week 6. In order to be considered for inclusion in the optimized intervention, intervention components must result in a 3-point decrease in T-score on the Patient-Reported Outcomes Measurement Information System (PROMIS)® Computer Adaptive Test (CAT) for depression between W0 and W6. T-scores have a range from 0 to 100, a mean of 50, and a standard deviation of 10. On this measure, higher scores indicate greater depressive symptoms (worse outcome).

SECONDARY OUTCOMES:
Change in Depressive Symptoms at follow-up | Baseline to Week 12
  The investigators will also evaluate change in depressive symptoms from Week 0 to Week 12 and Week 24 using the Patient-Reported Outcomes Measurement Information System (PROMIS)® Computer Adaptive Test (CAT) for depression. T-scores have a range from 0 to 100, a mean of 50, and a standard deviation of 10. On this measure, higher scores indicate greater depressive symptoms (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Karly M Murphy, PhD, Principal Investigator — East Carolina University
Locations (2):
- United States (2):
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data collected from participants in this study will be preserved and shared in alignment with best practices for open science. Data will be submitted to Dataverse, a free NIH Generalist Repository Ecosystem Initiative (https://dataverse.org/researchers).
Supporting Information: Study Protocol, ICF